CLINICAL TRIAL: NCT04726826
Title: Predictive Biomarkers of Mortality and Morbidity in Children Hospitalized for Acute Febrile Illness
Brief Title: Biomarkers of Mortality and Morbidity in Children Hospitalized With Fever
Status: Completed | Type: Observational
Sponsor: University of Alberta (Other)
Collaborators: University of Toronto (Other); Global Health Uganda LTD (Other)
Responsible Party: Sponsor
Other Study IDs: Pro00106489
Record Dates: First submitted 2021-01-19; First posted 2021-01-27 (Actual); Last update posted 2021-01-27 (Actual); Status verified 2021-01

CONDITIONS: Fever
Keywords: fever; child; biomarker
MeSH Terms: conditions — Fever | interventions — Diagnosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Serum and plasma obtained by venipuncture at hospital admission
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Diagnostic and prognostic biomarkers — Observational study of biomarkers predictive of morbidity and mortality in febrile children

SUMMARY:
The objective of this study is to identify clinically informative biomarkers of host defense pathways with potential utility as diagnostic and prognostic tools among children hospitalized with acute febrile illness in a resource-constrained sub-Saharan African setting.

The working hypothesis is that a panel of biomarkers, readily measurable from a peripheral blood sample, may serve as a clinically useful instrument to distinguish between common pediatric causes of fever, predict those children at greatest need of aggressive supportive care and/or adjunctive therapies, and identify those children at greatest risk of mortality. The use of objective and quantitative tools may facilitate the triage and clinical care of febrile children admitted to hospital in the sub-Saharan African context.

DETAILED DESCRIPTION:
For pediatric patients presenting to Jinja Regional Referral Hospital in whom admission to hospital is deemed necessary by an attending physician, the parent or guardian will be approached for consent to participate in the study. If granted, a small volume (1mL) of blood will be withdrawn for processing and storage. A RDT for malaria and whole blood lactate level will be performed at the bedside. Basic demographic and clinical data will be collected from the case admission record, and patients will be followed during their hospital admission. Possible outcomes will include: death, discharge without disability, discharge with disability, abscondment, and loss to follow-up. The length of stay among survivors will be recorded (excluding patients leaving against medical advice).

Serum samples will be shipped to the collaborating laboratory in Canada for analysis for biomarkers. ELISA-based commercially-available assays for biomarker levels will be used to quantify biomarker levels. In order to measure levels of 13 biomarkers from a plasma sample of 500uL or less, highly co-ordinated procedures with experienced technicians are required to perform the ELISA. Our laboratory in Canada has established protocols, experienced staff able to perform the testing, as well as equipment and reagents allowing the testing to be done efficiently. While it would be desirable to augment Ugandan capacity for biomarker testing, this would require significant investment of time and resources for training and testing, and may not be feasible in the context of this early study. If biomarkers can be identified that have clinical utility, laboratory capacity for ELISA measurement of levels should be developed or a simplified platform (e.g., lateral flow immunochromatographic test) should be developed.

Pneumonia and meningitis will be diagnosed clinically. A combination of tachypnea, respiratory distress (nasal flaring, intercostal and/or subcostal indrawing, or cyanosis) and characteristic findings on chest auscultation (asymmetrical air entry, crackles, dullness to percussion) will be used to make a clinical diagnosis of pneumonia. In our setting, chest x-ray is not available on site and radiographic confirmation will not be routinely available. Neck stiffness, positive Kernig's or Brudzinsky's signs, convulsions and coma will be used to make a diagnosis of meningitis. Where a lumbar puncture is performed, according to clinical judgment, the results will be used to complement clinical diagnosis. CSF pleiocytosis or a positive CSF culture for recognized pathogens will be used to support the diagnosis of meningitis.

ELIGIBILITY:
Inclusion Criteria:

1. Age 2 months to 5 years
2. History of fever within past 48 hours or axillary temperature >37.5°C
3. Hospital admission warranted based on clinician judgment
4. Consent to blood sampling and data collection

Exclusion Criteria:

1. Outside eligible age range
2. No history or objective evidence of fever
3. Diarrheal illness without other symptoms
4. Outpatient management
5. Denial of consent to participate in study

Ages: 2 Months to 5 Years | Sex: All
Age Groups: Child
Study Population: The choice of the age range for this study is as follows. Children under 5 represent a vulnerable group, in whom infectious diseases play a major role as contributors to overall mortality. Children under 2 months of age (the neonatal group) represent a unique population with different infectious risks and are therefore outside the scope of our current study.
  The reason for exclusion of isolated diarrheal illness is that dehydration, acidosis and electrolyte imbalances are the proximal causes of mortality, rather than activation of host defense pathways with excessive inflammation and endothelial activation. Host biomarkers are therefore not expected to predict mortality with the same accuracy in diarrhea syndromes.
Sampling Method: Non-Probability Sample
Enrollment: 2500 (Actual)
Dates: Start 2012-02-01 (Actual); Primary Completion 2013-09-15 (Actual); Study Completion 2013-09-15 (Actual)

PRIMARY OUTCOMES:
Mortality | through study completion, an average of 1 week
  in-hospital mortality

SECONDARY OUTCOMES:
Hospital length of stay | through study completion, an average of 1 week
  time from admission to discharge
Lambarene organ dysfunction score (LODS), a composite clinical severity score | evaluated at admission
  clinical severity score
Signs of Inflammation in Children that Kill (SICK), a composite clinical severity score | evaluated at admission
  clinical severity score

CONTACTS AND LOCATIONS:
Overall Officials: Michael T Hawkes, MD, PhD, Principal Investigator — University of Alberta
Locations (1):
- Jinja Regional Referral Hospital, Jinja, Uganda

IPD SHARING:
Plan to Share IPD: Yes
Data will be shared upon reasonable request to study prinicipal investigator.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: 10 years
Access Criteria: Upon reasonable request to study principal investigator.

REFERENCES:
- [Derived] McDonald CR, Leligdowicz A, Conroy AL, Weckman AM, Richard-Greenblatt M, Ngai M, Erice C, Zhong K, Namasopo S, Opoka RO, Hawkes MT, Kain KC. Immune and endothelial activation markers and risk stratification of childhood pneumonia in Uganda: A secondary analysis of a prospective cohort study. PLoS Med. 2022 Jul 13;19(7):e1004057. doi: 10.1371/journal.pmed.1004057. eCollection 2022 Jul. PMID 35830474